CLINICAL TRIAL: NCT06458894
Title: Research on Building and Application of Internet-based Home Pre-rehabilitation Model for Lung Surgery Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY-2024-102
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- There were no interventions (Other): Give guidance on respiratory function exercise
  Interventions: Behavioral: Prerehabilitation
- Prerehabilitation (Other): Give guidance on respiratory function exercise
  Interventions: Behavioral: Prerehabilitation

INTERVENTIONS:
Behavioral: Prerehabilitation — Home prerehabilitation was performed on the basis of routine preoperative preparation
  Other Names: ulmonary function

SUMMARY:
This study, based on the Internet platform, involving family caregivers in preoperative management, not only promotes patient compliance with preoperative rehabilitation exercise, but also provides multi-way rehabilitation measures for elderly patients with limited mobility or medical difficulties, and also provides new ideas for other specialties。

DETAILED DESCRIPTION:
This study using a randomized controlled trial, 100 patients that meet the inclusion criteria are divided into experimental group and control group, experimental group adopts routine nursing measures, intervention group for preoperative family rehabilitation training, intervention for 2 weeks, observe the first after surgery, lung function index, chest catheterization days, postoperative hospital stay and medical expenses.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years old; 2. A preliminary diagnosis of pulmonary结节 or lung tumor by chest CT; 3. Planning to undergo thoracoscopic lung resection surgery; 4. Voluntary participation of patients.

Exclusion Criteria:

1. Patients with severe condition who cannot tolerate pre-rehabilitation training; 2. Patients with consciousness disorder or mental abnormalities who cannot cooperate with pre-rehabilitation training; 3. Patients who cannot complete questionnaire filling out due to visual, auditory, or intellectual impairment, etc.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Time to the first ambulation after surgery | 3 Weeks after intervention
  Patients can complete the time of walking at the bed, and unplanned extubation
Dwelling time of chest drain and chest drainage flow | Two days after the intervention
  The duration of the postoperative chest drain and the chest on postoperative day 1 and postoperative day 2 were recorded Lead the flow

SECONDARY OUTCOMES:
Lung function index | 30 Days after intervention
  Pulmonary function test was performed with the pulmonary function detector on the day of the patient and 30 days after surgery Guide the patient to do inhale or exhale with maximum effort, make three consecutive measurements, and record the best results, including Forced expiratory volume at second 1

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No